CLINICAL TRIAL: NCT00859599
Title: Monochromatic Phototherapy on Diabetic Foot Ulcers. A Twenty Weeks Prospective, Randomised, Double Blind, Multi-centre, Placebo Controlled Study
Brief Title: Monochromatic Phototherapy on Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biolight AB (Industry)
Responsible Party: Hans Johansson, Manager Clinical Trials And Product Manager Wound, Biolight AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BL-039; H15:321/2008
Record Dates: First submitted 2009-02-27; First posted 2009-03-11 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Foot Ulcers
Keywords: Monochromatic Phototherapy; Diabetic Foot Ulcers; Wound healing; Bacterial colonisation
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): At the study start, the patient will be given a subject number according to a fixed randomisation list. The investigator/study nurse will be instructed to log in at the Biolight® website to get the patient-number and treatment code, with the information which treatment model (i.e. marked A & B, E & F, X & Y) the randomised patient shall receive.
  Up to 44 monochromatic Phototherapy treatment sessions (Biolight® or placebo) will be given, additional to standard care treatment. The treatment session schedule compromise of three times weekly during the first four weeks and twice weekly during the following weeks or until the ulcer is completely healed.
  Interventions: Device: Monochromatic phototherapy, Biolight®; Device: Monochromatic phototherapy
- 2 (Placebo Comparator): At the study start, the patient will be given a subject number according to a fixed randomisation list. The investigator/study nurse will be instructed to log in at the Biolight® website to get the patient-number and treatment code, with the information which treatment model (i.e. marked A & B, E & F, X & Y) the randomised patient shall receive.
  Up to 44 monochromatic Phototherapy treatment sessions (Biolight® or placebo) will be given, additional to standard care treatment. The treatment session schedule compromise of three times weekly during the first four weeks and twice weekly during the following weeks or until the ulcer is completely healed.
  Interventions: Device: Monochromatic phototherapy, Biolight®; Device: Monochromatic phototherapy

INTERVENTIONS:
Device: Monochromatic phototherapy, Biolight® — Monochromatic phototherapy (Biolight®) will be given locally, additional to standard care, three times weekly during the first four weeks and twice weekly the following sixteen weeks or until the ulcer is completely healed, according to a pre-determined treatment plan.
  Other Names: Biolight® Care Device (BCD); Biolight® Wound Care Device (WCD); Monochromatic Light Therapy; Monochromatic phototherapy
Device: Monochromatic phototherapy — Monochromatic phototherapy (Biolight®) will be given locally, additional to standard care, three times weekly during the first four weeks and twice weekly the following sixteen weeks or until the ulcer is completely healed, according to a pre-determined treatment plan.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of monochromatic phototherapy (Biolight®) on foot ulcers in diabetic patients, in comparison of placebo phototherapy as a complementary to standard diabetic foot ulcer therapy.

The study initiated with a four week long Run In Period to eliminate spontaneous healing ulcer to be included. Treatment with monochromatic phototherapy (Biolight® or placebo) will be given locally, additional to standard care, three times weekly during the first four weeks and twice weekly the following sixteen weeks or until the ulcer is completely healed, according to a pre-determined treatment plan. The area of the ulcer will be measured once weekly for 20 weeks or until the ulcer is completely healed.

DETAILED DESCRIPTION:
Description of Biolight® Therapy and device The therapy works by applying, for each indication, a specific combination of pulsating monochromatic light to specific areas of the body. The therapy is non-invasive, non-thermal, and based on the effects of pulsed monochromatic light in the visible or near-visible spectrum.

The Biolight® Therapy - mechanism of action Light is a pre-requisite for most living organisms, and human being have learnt to use light in many different situations, not least in health care, where light is widely used in various therapeutic contexts every day. X-ray is used as an investigational tool. In treating skin diseases, such as psoriasis, we use UV radiation. Laser has been successful, both in surgery and for pain relief, and white light treatment is recommended in seasonal depressions

Light is in fact electromagnetic radiation using various wavelengths. These wavelengths are perceived as different colours. Red and violet light consist of long and shorter wavelength respectively. Light consisting of all the wavelengths is perceived as white. There is an electromagnetic field in light containing energy, which can be used in different treatment situations.

In the healing process of wounded tissue basal components need access to energy and oxygen. If the amount of energy is insufficient, the healing process is retarded. By the use of monochromatic light, having a predetermined energy level and a specific wavelength, we can contribute to the expected amount of energy demand. Applied at a chosen pulse frequency and for a carefully calculated period of time, the wounded cells are provided with energy, increasing their activity as well as the oxygen supply in the damaged area. That may promote a faster healing.

The Biolight Therapy is suggested to shorten treatment time and reduce treatment costs and to improve quality of life. This non-invasive treatment is thought to be complementary to traditional therapies. The method is simple, painless and without known side effects.

The Biolight Care Device The Biolight® Care Device is a CE-marked medical device certified in accordance with the Medical Device Directive (MDD; 93/42/EEC), with the size of the palm of the hand.

The device contains 30 diodes emitting infrared light at 956 nm and also 80 diodes emitting red light at 637 nm. Infrared and red pulsed monochromatic light are used in a unique triple-stepped sequence. Infrared light, with an irradiance of ~55 W/m2, is combined with red light, with an irradiance of ~21 W/m2. Using a duty cycle of 80%, both infrared and red light are pulsed at the following frequencies during the first week: infrared/red 78 Hz, infrared/red 702 Hz, infrared/red 8572,2Hz and from the second week: infrared/red 15,6 Hz, infrared/red 287 Hz, infrared/red124 Hz. The choice of pulse frequencies and wavelengths are based on earlier observations in both in-vitro and in-vivo studies. The equipment for both monochromatic phototherapy and placebo (no irradiance output from the diodes) is identical in appearance.

Previous studies - light therapy Treatment with pulsed electromagnetic fields for 40 minutes improves micro vascular perfusion of the skin (1). In a literature overview from 1965 to 2003 on low-laser therapy for wound healing, focusing on both in vitro models and in vivo animal and human studies, some studies reported increased cell proliferation and collagen production; improvements in surgical wound healing were found in a rodent model; and, in humans, beneficial effects on superficial wound healing found in small case series have not been replicated in larger studies (2). In none of the reviewed studies was the exact mechanism of photo thermal, photochemical or photomechanical action, reported.

The precise mode of action of low-laser therapy on wound healing is still unknown (2). In a meta-analytic study of 34 peer-reviewed papers on the efficacy of low-power lasers in tissue repair, a positive effect was shown on collagen formation, rate of healing, tensile strength, and time needed for wound closure (3). In an experimental study on pressure ulcers in mice, a significant positive effect was shown on wound healing after treatment with low-laser therapy and this effect was independent of the temperature on the skin surface (4). In a systematic review of the effects of low-level laser therapy on wound healing in cell studies and animal model experiments by Lucas et al. (5), the 36 included studies contained 49 outcome parameters, of which 30 reported the positive effect of laser irradiation and 19 did not. The methodological quality of many studies was poor, and in-depth analysis of the studies with the highest methodological quality scores showed no significant pooled effect in favour of treatment (5).

A study of 20 spinal cord-injured patients with 22 pressure ulcers showed faster healing with a combination of ultrasound/ultraviolet-C and laser treatment, compared with nursing care alone (6). In a prospective, observer-blinded, multicenter randomized clinical study on the efficacy of low-level laser therapy in 86 patients with stage III decubitus ulcers, no evidence was found that justified the use of low-level laser therapy (7).

Previous studies - Biolight® A double-blind randomized placebo-controlled study on pressure ulcer in elderly patients showed a statistically significant difference between patients treated with monochromatic pulsating light (Biolight®) or placebo together with standard care. This study was conducted on 163 patients as a multi-centre study at 9 centres in Sweden and Denmark (8, 9). The mean normalised reduction in pressure ulcer size at week 12 was 0.79 for the phototherapy group and 0.50 for the placebo group (95 % CI 0.01-0.53; p=0.039). No serious side effects were noted. The conclusion was that monochromatic pulsating light fastened healing in grade II pressure ulcers in elderly patients.

A sub group analysis for the patient with diabetic foot ulcer in the above study showed a strong tendency to improved healing (diff 71.3%).

A controlled, randomised, open study on the effect of Biolight® phototherapy in comparison to conventional treatment in 74 patients with grade II or III chronic pressure ulcers was conducted at Huddinge hospital (10). This study showed a statistically significant decreased time to healing, in the phototherapy treated group compared with the control group.

A clinical study of 26 elderly patients with decubitus ulcers showed that monochromatic phototherapy, Biolight®, had an effect on the microcirculation in the edge of the decubitus ulcer with an increase of the oxygen supply to the tissue. (12).

Two in-vitro studies on the growth of skin fibroblast cells, using monochromatic phototherapy showed that the two wavelengths and the low and high pulse frequencies used in the Biolight® Wound Care program significantly influenced skin fibroblast cell growth (personal communication Kratz & Huss Karolinska Institute, Stockholm, Sweden).

In an animal study (exposure 5 times a week during a 2-week period), with similar equipment and similar infrared and red light exposure as in the present study, no adverse effect was found (11).

Study population Diabetic patients with foot ulcers will be randomised to active phototherapeutic treatment plus standard care treatment or placebo phototherapeutic treatment plus standard care for diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Wagner grade 1-2 (superficial or deep ulcer)
* Size of ulcer 1 -25 cm2
* Localisation of the ulcer below the ankle
* Systolic ankle blood pressure >80 mmHg or
* Systolic toe blood pressure >45 mmHg equal to and higher than or only
* Type 1 or II diabetes - Previously known diabetes according to WHO criteria
* HbA1c <12
* > 18 year
* Willing and able to fulfil the study requirements
* Written informed consent

Exclusion Criteria:

* Earlier participation in this study
* Life-threatening malignancy
* Systemic, oral use of corticosteroid preparations (> 7.5 mg Prednisolon)
* Immunosuppressive treatment such as cytostatic drugs and TNF-antagonists
* Kidney insufficiency (Creatinine >250 micromol/l)
* Clinical signs of infections
* Antibiotic treatment the last two weeks
* Suspected venous genesis
* More than two ulcers per foot
* Wagner grade 3-5
* Location of ulcers making treatment or evaluation not feasible
* Photosensitivity or other sensitivity to electromagnetic radiation
* Pregnancy or breastfeeding
* Participation in any clinical study the last three month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who completely healed and time to 100% wound reduction. | 24 weeks

SECONDARY OUTCOMES:
Time to 50% wound reduction, Subjects with increased ulcer and/or wound reduction less than 20%, Wound status, Elimination of gram-positive and anaerobic bacteria from the wound, Hospitalization caused of foot ulcer, Presence and level of amputation | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Apelqvist, M.D., Ph.D., Principal Investigator — Malmö University Hospital, Department of Endocrinology
Locations (7):
- Sweden (7):
  - Department of Medicine, Ängelholm, Skåne County
  - Frölunda Specialistsjukhus, Gothenburg
  - Regional Hospital, Halmstad, Halmstad
  - Karolinska University Hospital, Huddinge
  - Lund University Hospital, Lund
  - Malmö University Hospital, Malmo
  - Uddevalla Hospital, Uddevalla